CLINICAL TRIAL: NCT03934190
Title: Inner Nuclear Macular Microcyst is a Risk Factor for Macular Cystoid Changes After Phacoemulsification in Eyes With Previous Vitrectomy and Macular Pucker Removal
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, San Ni Chen, Director of Department of Ophthalmology, Changhua Christian Hospital
Other Study IDs: 141012
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Macular Pucker; Macular Cyst
Keywords: macular edema; pseudophakic cystoid macular edema; macular pucker; internal limiting membrane peeling; pars plana vitrectomy
MeSH Terms: conditions — Epiretinal Membrane; Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the visual acuity, macular thickness, morphological changes after cataract surgery in eyes with previous vitrectomy for macular pucker. Associated risk factors were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients had macular pucker surgery before cataract surgery.
* Follow up over 1 year.

Exclusion Criteria:

* Patients had any surgical complications such as posterior capsule rupture, vitreous loss, prolapse through the wound or iris trauma
* Patients had diabetes mellitus.
* Patients had uveitis or other inflammatory eye disease.
* Patients had history of retinal vein occlusion.
* Patients had retinal detachment; or previous vitrectomy for a disease other than macular pucker.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The general medical history of the patients was evaluated preoperatively. Comprehensive ophthalmological examinations including BCVA measurements and funduscopic examinations were performed at each visit. SD-OCT (Cirrus HD-OCT, Carl Zeiss Meditec, Dublin, CA) was used to measure the central macular thickness (CMT) and structural changes preoperatively, and at 1 day, 1 week, 1 month, 3 months, 6 months and 1 year postoperatively
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Wilcoxon Signed-Rank test | 1 day, 1 week, 1 month, 3 months, 6 months and 1 year
  A statistical comparison of average of different time point

SECONDARY OUTCOMES:
visual acuity | 1 day, 1 week, 1 month, 3 months, 6 months and 1 year
  visual acuity change in logMAR in different time point

CONTACTS AND LOCATIONS:
Overall Officials: San-Ni Chen, MD, Principal Investigator — Changhua Christian Hospital